CLINICAL TRIAL: NCT07091799
Title: Interest of Measuring P2X4 Receptors on Blood Monocytes as a Diagnostic Marker in Amyotrophic Lateral Sclerosis: P2X4 as a Diagnostic Biomarker for ALS
Acronym: PALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2024/82
Record Dates: First submitted 2025-06-25; First posted 2025-07-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis &Amp; Other Neuromuscular Disorders
Keywords: P2X4; diagnostic biomarker; purinergic pathway
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALS patient (Experimental): During the inclusion visit on D0, which will take place during a consultation or a hospitalization scheduled as part of the standard of care, patients will be informed about the protocol and their informed consent will be obtained.
  A neurological clinical examination will be performed, the ALSFRS-R score will be evaluated, as well as respiratory functional explorations and a standard biology assessment. As part of the research, an additional blood sample will be taken.
  For ALS patients, a follow-up visit will be performed at 6 months as part of their follow-up consultation at the ALS center. The same examinations as on D0 will be done.
  Interventions: Diagnostic Test: P2X4 receptors in blood samples
- Standard : healthy subjects (Other): During the inclusion visit on D0, which will take place during a consultation or a hospitalization scheduled as part of the standard of care. A neurological clinical examination will be performed, the ALSFRS-R score will be evaluated, as well as respiratory functional explorations and a standard biology assessment. As part of the research, an additional blood sample will be taken.
  For healthy subjects, a follow-up visit will be performed at 6 months. The same examinations as on D0 will be done.
  Interventions: Diagnostic Test: P2X4 receptors in blood samples

INTERVENTIONS:
Diagnostic Test: P2X4 receptors in blood samples — This is an interventional study designed to assay P2X4 receptors in blood samples from ALS patients and healthy volunteers by comparing the mean levels of P2X4 expression.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is the most common form of motor neuron disease and is characterized by the degeneration of motor neurons leading to progressive paralysis and death within 3 to 5 years after diagnosis. To date, no key mechanism had been identified. Our associated laboratory has identified the P2X4 purinergic pathway that appears to be involved in the pathogenesis of ALS. Our goal is to verify these results at the human level in order to have a proof of concept of P2X4's role as a biomarker of the disease.

ELIGIBILITY:
Inclusion Criteria:

* For ALS group: Person presenting a probable or confirmed diagnosis of ALS according to the criteria of EI Escorial.
* Adult.
* Person affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant or by a third person (in case of physical incapacity of the participant), after information on the study.

Exclusion Criteria:

* People undergoing immunosuppressive or corticosteroid treatments.
* Participation in a research protocol with an experimental treatment.
* People placed under guardianship, curatorship or legal protection.
* For healthy volunteer, people directly related to the patient (siblings, descendants and ancestry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Expression of P2X4 receptor | 6 months after Day 0
  Compare expression of P2X4 receptor in ALS patients versus healthy subjects to demonstrate its role as a clinical biomarker of ALS. Comparison will be obtained by labeling and flow cytometer analysis of circulating monocytes.

SECONDARY OUTCOMES:
Diagnostic performance | 6 months after Day 0
  Evaluate the diagnostic performances of P2X4 receptor assay for the diagnosis of ALS, thanks to sensitivity and specificity of this P2X4 receptor assay
Prognostic performances | 6 months after Day 0
  Evaluate prognostic performances of P2X4 receptor assay for the diagnosis of ALS, thanks to sensitivity and specificity of this P2X4 receptor assay
P2X4 receptor levels evolution | 6 months after Day 0
  Describe evolution of P2X4 receptor levels with a new sample at 6 months in the same patients, thanks to the difference in P2X4 receptor expression average in the same ALS patient
Levels of P2X4 receptors between patients with familial or sporadic ALS. | 6 months after Day 0
  Compare expression levels of P2X4 receptors between patients with familial or sporadic ALS, thanks to the difference in P2X4 receptor expression average
P2X4 receptor levels of patients with a SOD1 mutation treated with anti-SOD1antisense | 6 months after Day 0
  Compare surface P2X4 receptor levels of patients with a SOD1 mutation treated with anti-SOD1 antisense (Qalsody®, TOFERSEN), thanks to the difference in P2X4 receptor expression average

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No